CLINICAL TRIAL: NCT04409808
Title: IRIS Alfa Clinical Trial. A Safety Study of a Prototype of a New Vitrectomy Device.
Brief Title: IRIS Alfa Clinical Trial A Monocentric, Academic Clinical Trial Safety Study of a Prototype of a New Vitrectomy Device.
Acronym: IRIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because a device deficiency that occured in the Iris vitrectomy system (Alfa version)
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S62660
Record Dates: First submitted 2020-05-05; First posted 2020-06-01 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2021-09

CONDITIONS: Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRIS vitrectomy device (Experimental): all subjects in this study are in the experimental treatment arm and vitrectomy by use of prototype IRIS vitrectomy device
  Interventions: Device: IRIS

INTERVENTIONS:
Device: IRIS — prototype IRIS vitrectomy device.

SUMMARY:
To perform a safety study on the prototype IRIS vitrectomy device.

DETAILED DESCRIPTION:
to determine the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are scheduled for vitrectomy surgery, regardless of the indication
* Both vitrectomy-only and combined phaco-vitrectomy surgeries
* Primary or repeat vitrectomy
* General or local anesthesia, or combination
* All ages
* Informed consent (from parents in patients <18 years old)

Exclusion Criteria:

* Unable to obtain informed consent from patient (or from parents in children)
* No post-operative 8 week visit is anticipated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
incidence of intra-operative adverse events that determine the safety of the surgery | Intraoperative (surgery day)
  complications VTX: iatrogenic tear, lens touch, choroidal/subretinal/vitreous hemorrhage, infusion suprachoroidal, iatrogenic retina trauma, posterior capsule tear, corneal eptihelial damage, hyphema, corneal edema, iris trauma, nucleus fragment in vitreous, posterior capsule tear, retinal incarceration, zonulae rupture with vitreous prolapse, subretinal PFCL, suprachoroidal silicone oil, zonulae dialysis, lens exchange required, other IOL problem

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PHd MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No